CLINICAL TRIAL: NCT03994640
Title: Myorelaxant Effect of Cannabis Cream Topical Skin Application in Patients With Temporomandibular Disorders: a Randomized, Double-blind Study
Brief Title: Myorelaxant Effect of Cannabis Cream Topical Skin Application in Patients With TMD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Aleksandra Nitecka-Buchta, Principal Investigator, Medical University of Silesia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Silesian UM Cannabis
Record Dates: First submitted 2019-06-17; First posted 2019-06-21 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Temporomandibular Disorder; Myofascial Pain; Cannabis; Electromyography
Keywords: temporomandibular disorder; Cannabis; Electromyography; Masticatory muscles; Topical application
MeSH Terms: conditions — Temporomandibular Joint Disorders; Marijuana Abuse

STUDY DESIGN:
Intervention Model Description: two groups parallel study: experimental and control group
Who Masked: Participant, Care Provider
Masking Description: double blind study: for patients and researchers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cannabis cream (Experimental): Cannabis cream topical skin application in experimental group
  Interventions: Combination Product: Cannabis Cream
- Placebo cream (Placebo Comparator): Placebo cream topical skin application in control group
  Interventions: Combination Product: Placebo Cream

INTERVENTIONS:
Combination Product: Cannabis Cream — Topical, bilateral skin application of cannabis cream with self-massage of masseter muscles
  Other Names: Cannabis cream topical skin application
  Arms: Cannabis cream
Combination Product: Placebo Cream — Topical, bilteral skin application of placebo cream with self-massage of masseter muscles
  Other Names: Placeo cream topical skin application
  Arms: Placebo cream

SUMMARY:
Evaluation of myorelaxant effect of cannabis cream.compared to placebo cream in topical skin application in patients with TMD

DETAILED DESCRIPTION:
Cannabis sativa has a very wide application in various fields of medicine. In patients with temporomandibular disorder, especially with myofascial pain of masticatory muscles there is a special need to seek an effective pain therapy and muscle relaxing methods. Patients with TMD suffer from chronic pain and depression, cannabis topical skin application therapy seems promising in that field. Patients attending The Department of TMD in Zabrze, Polska were randomly divided into two groups: experimental and placebo. sEMG activity values were compared during 14 days therapy with cream. Positive results were obtained confirming the efficacy of the cannabis cream used in the study, compared to placebo.

ELIGIBILITY:
The inclusion criteria were as follows:

1. Patient agreement to participate into the research study
2. Age ≥22 and ≤ 27
3. Good general health,
4. Temporomandibular disorder-positive RDC/TMD examination for group Ia and Ib
5. Presence of all teeth (with the exception of the third molars)

The exclusion criteria were:

1. Cannabis cream/ placebo cream allergy
2. Hypersensitivity to substances to be used in the study
3. Skin wounds with skin surface discontinuation
4. Addiction to cannabis
5. Patients being treated with analgesic drugs and/or drugs that affect muscle function
6. Fixed or removable dental prosthesis
7. Disease or autoimmune disorder associated with generalized muscular tension

Ages: 22 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Reduction of sEMG activity of masseter muscle | 14 days
  Reduction in masseter muscle electromyographic activity

CONTACTS AND LOCATIONS:
Locations (1):
- Department of TMD Silesian Medical University, Zabrze, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vaney C, Heinzel-Gutenbrunner M, Jobin P, Tschopp F, Gattlen B, Hagen U, Schnelle M, Reif M. Efficacy, safety and tolerability of an orally administered cannabis extract in the treatment of spasticity in patients with multiple sclerosis: a randomized, double-blind, placebo-controlled, crossover study. Mult Scler. 2004 Aug;10(4):417-24. doi: 10.1191/1352458504ms1048oa. PMID 15327040
- [Background] Koppel BS, Brust JC, Fife T, Bronstein J, Youssof S, Gronseth G, Gloss D. Systematic review: efficacy and safety of medical marijuana in selected neurologic disorders [RETIRED]: report of the Guideline Development Subcommittee of the American Academy of Neurology. Neurology. 2014 Apr 29;82(17):1556-63. doi: 10.1212/WNL.0000000000000363. PMID 24778283
- [Background] Schiffman E, Ohrbach R, Truelove E, Look J, Anderson G, Goulet JP, List T, Svensson P, Gonzalez Y, Lobbezoo F, Michelotti A, Brooks SL, Ceusters W, Drangsholt M, Ettlin D, Gaul C, Goldberg LJ, Haythornthwaite JA, Hollender L, Jensen R, John MT, De Laat A, de Leeuw R, Maixner W, van der Meulen M, Murray GM, Nixdorf DR, Palla S, Petersson A, Pionchon P, Smith B, Visscher CM, Zakrzewska J, Dworkin SF; International RDC/TMD Consortium Network, International association for Dental Research; Orofacial Pain Special Interest Group, International Association for the Study of Pain. Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) for Clinical and Research Applications: recommendations of the International RDC/TMD Consortium Network* and Orofacial Pain Special Interest Groupdagger. J Oral Facial Pain Headache. 2014 Winter;28(1):6-27. doi: 10.11607/jop.1151. PMID 24482784